CLINICAL TRIAL: NCT04094077
Title: A Phase II Study Evaluating AGuIX® Nanoparticles in Combination With Stereotactic Radiation for Oligo Brain Metastases.
Brief Title: Evaluating AGuIX® Nanoparticles in Combination With Stereotactic Radiation for Brain Metastases
Acronym: NANOSTEREO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped after a negative result delivred by the CPP for a substancial modification of the protocol
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ET18-270 NANOSTEREO
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Brain Metastases
Keywords: Stereotactic Radiation; Nanoparticles
MeSH Terms: conditions — Brain Neoplasms | interventions — AGuIX

STUDY DESIGN:
Intervention Model Description: This study is a paucicentric, single arm Phase II trial conducted according to a single stage Fleming-A'Hern design and aiming to evaluate the efficacy of AGuIX® during FSRT of brain metastasis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aguix + Stereotactic Radiation (Experimental)
  Interventions: Drug: AGuIX

INTERVENTIONS:
Drug: AGuIX — 2 IV injections (100 mg/Kg/injection) at day 4 and day 8 + Strereotactic Radiation from day 8 to day 15 as per standard practice.

SUMMARY:
This study evaluates the clinical impact of AGuIX® nanoparticles in combination with Fractionated Stereotactic Radiation in oligo brain metastases.

DETAILED DESCRIPTION:
AGuIX® (Activation and Guidance of Irradiation by X-ray, NH TherAguix) are Gadolinium chelated polysiloxane based nanoparticles with Magnetic Resonance contrast properties, able to accumulate in the tumor through the enhanced permeability and retention effect and sufficiently small (sub-5 nm diameter) to allow for renal clearance.

AGuIX® nanomedicine can be used as:

* Positive contrast agent for Magnetic Resonance Imaging (MRI). It displays higher efficacy than commercial contrast agents and so it can be used to delineate precisely the tumors.
* A booster of Radiotherapy during the radiotherapy protocol, after the localization of the tumor.

This is permitted by the high radiosensitizing potential of AGuIX® that allows a local increase of efficacy of X-ray damages. French and international groups have demonstrated the radiosensitizer effect of AGuIX® to improve the efficacy of radiotherapy.

Thanks to a difference in porosity between the vascular networks, AGuIX® penetrates and resides in tumor tissues, but not in healthy tissues.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged of at least 18 years on day of signing informed consent.
* Histologically-confirmed diagnosis of any histological type of solid tumors, excluding primary central nervous system (CNS) tumors.
* Radiological evidence by MRI : At least one and a maximum of 5 brain metastases, and at least one brain lesion with a longest diameter ≥ 2 cm and eligible for FSRT.
* Patient without progression on extracranial disease documented by radiological assessment as per RECIST v1.1 within 4 weeks before inclusion.
* For patients treated with a systemic anti-cancer therapy: a minimal 2-week washout period is required from the date of last systemic treatment administration to Day 1, except for hormonal agents.
* ECOG Performance Status (PS) ≤2.
* Absolute neutrophil count (ANC) ≥ 1.0 G/L, Platelets ≥ 75 G/L, Hemoglobin ≥ 8 g/dL, Serum creatinine OR Creatinine clearance according to CKD-EPI ≤ 1.5 x Upper Limit of Normal (ULN) OR ≥ 50 mL/min/1.73m2, ASAT and ALAT ≤ 3 x ULN (or ≤ 5.0 ULN in case of liver metastasis or hepatic infiltration),INR and Activated Partial Thromboplastin Time (aPTT) ≤1.5 x ULN.
* Women of child-bearing potential must have a negative serum pregnancy test at screening and must agree to use 2 effective forms of contraception from the time of the negative pregnancy test up to 3 months after the last dose of the study drug.
* Fertile men must agree to use contraceptive measures up to 3 months after the last dose of study drug.
* Patients who understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Prior local treatment with radiotherapy (whole / partial brain or stereotactic radiosurgery) or surgical resection of brain lesions.
* Patient participating to another clinical trial with an investigational agent.
* Patients who have not recovered from significant adverse events (i.e. Grade > 2 AE according to NCI CTCAE v5.0) due to prior treatment with anti-cancer agents with exception of any Grade alopecia or lab values presented in inclusion criteria.
* Contra-indication for MRI enhanced with gadolinium (e.g. cardiac pacemaker, implanted defibrillator, certain cardiac valve replacements, certain metal implants).
* Patients who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Rate of local control | 1 year
  The primary endpoint is the rate of local control defined as the proportion of patients with a complete response, a partial response or a stable disease. Response of Brain lesion will be evaluated using the RECIST classifications with partial response (PR, > 30% decrease in longest diameter), stable disease (SD <30% decrease and <20% increase in longest diameter), progressive disease (PD > 20% increase in longest diameter) and Complete response (CR) (complete disappearance of the brain lesion).

SECONDARY OUTCOMES:
Distant Brain failure | 6 month and at 1 year
  Distant Brain failure is defined as the presence of new brain metastases or leptomeningeal enhancement outside the irradiated volume.
Time to brain relapse | 6 month and 1 year
  The event of interest will be the local progression on any irradiated lesion.
Tumor target volume | 4 days
  The Tumor target volume agreement is the comparison between both the MRI images with AGuIX® and Gd-chelates. It is defined as the correlation between the irradiation volume calculated based on the MRI before nanoparticles injection and the volume calculated after nanoparticles injection.
Brain lesion 3-D volume variation | 45 days and 3 month
  Brain lesion 3-D volume variation will be analysed using volumetric T1 post-gadolinium MRI.
Adverse events | From Day 1 to Day 45
  The assessment of safety will be based mainly on the frequency of adverse events based on the common toxicity criteria (CTCAE-V5.0) grade.
FACT-Br | 45 days, 3 month, 6 month, 9 month and 12 month
  The FACT-Br consists of a general version (FACT-G) and a brain subscale (BRCS). The FACT-G consist of 27 questions with 4 domains assessing physical well-being (score range: 0-28), social/family well-being (score range: 0-28), emotional well-being (score range: 0-24) and functional well-being (score range: 0-28). The BRCs is a 23-item questionnaire related to neurological concerns that provides an additional set of disease-specific questions pertaining to brain neoplasms (score range: 0-92). The FACT-Br total score is the sum of the FACT-G total score and the BrCS score. Positive change scores indicate improved quality of life.
MMSE | 45 days, 3 month, 6 month, 9 month and 12 month
  The MMSE is an 11-item measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall and language. The minimum score is 0 and the maximum score is 30 with higher MMSE scores indicating better cognition.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice